CLINICAL TRIAL: NCT03683290
Title: Efficiency of Modulation Contrast Microscopy Image Analysis as a Predictive Tool for Human Oocyte Quality
Brief Title: Modulation Contrast Microscopy Imaging for Oocyte Quality Assessment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Center for Reproductive an Genetic Health (Industry)
Collaborators: University College, London (Other)
Responsible Party: Principal Investigator, Xavier Vinals Gonzalez, Principal investigator, Center for Reproductive an Genetic Health
Other Study IDs: oocyte_imaging_2018
Record Dates: First submitted 2018-09-18; First posted 2018-09-25 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Oocyte Competence
Keywords: Oocyte; Embryo; Development; Pregnancy; Competence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 40 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Image acquisition and analysis — Oocyte image obtention and analysis prior to intracytoplasmic sperm injection

SUMMARY:
The present study aims to describe novel non-invasive parameters related to the competence of female reproductive cells (oocytes). In a fertility unit, human reproductive cells and embryos are subjected to different imaging technologies. Images can easily be obtained without disturbing the microenvironment during different standard procedures. Turning images into quantifiable data might provide a further understanding on oocyte behavior and performance in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Intracytoplasmic sperm injection
* Embryo culture with subsequent fresh embryo transfer

Exclusion Criteria:

- Conventional IVF

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Registered patients at The Centre for Reproductive and Genetic Health
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Implantation | 6 weeks gestation
  Number of gestational sacs seen on ultrasound scan

SECONDARY OUTCOMES:
Live Birth | 40 weeks gestation
  Baby to be born after embryo transfer
Fertilisation | 17 ± 1 hours post insemination
  Appearance of two pronucleii after insemination
Embryo quality clevage | 68 ± 1 hours post insemination
  Quality after three days of culture
Embryo quality Blastocyst | 116 ±2 hours post insemination
  Quality at the blastocyst stage
Euploidy | 2-3 weeks post insemination
  Number of chromosomes (if available, after PGT-A)
Nuclear maturity | 36-41 post hCG
  Presence of meiotic spindle (if available, PolScope)

CONTACTS AND LOCATIONS:
Overall Officials: Sioban SenGupta, Study Chair — Institute for Women's Health (UCL)
Locations (1):
- Centre for Reproductive and Genetics Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be collected and analysed internally. Results will be available (if published) in a scientific journal.